CLINICAL TRIAL: NCT07292012
Title: Efficacy of MIrikizumab to Achieve Transmural Healing in patiENTs With Crohn's Disease : EMINENT-CD
Brief Title: Efficacy of MIrikizumab to Achieve Transmural Healing in patiENTs With Crohn's Disease
Acronym: EMINENT-CD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GETAID-2025-02; 2025-521889-95-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease (CD)
Keywords: crohn's disease; transmural healing; mirikizumab
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mirikizumab treatment (Experimental): Mirikizumab will be used as scheduled in the drug label: induction with IV infusions (900 mg) at week 0, week 4 and week 8.
  For clinical responders: SC injections (300 mg) at W12 and every 4 weeks For clinical non-responders: SC injections (300 mg) at W12 and every 4 weeks
  Interventions: Drug: Mirikizumab - IV; Drug: Mirikizumab - SC

INTERVENTIONS:
Drug: Mirikizumab - IV — Mirikizumab induction with IV infusions (900 mg) at week 0, week 4 and week 8.
Drug: Mirikizumab - SC — SC injections (300 mg) at W12 and every 4 weeks For clinical responders and non-responders

SUMMARY:
Efficacy of Mirikizumab to achieve transmural healing in patients with Crohn's Disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD
* ≥ 18 to ≤ 75 years-old
* Symptomatic CD according to PRO-2 (stool > 3 or abdominal pain score > 1)
* Transmural inflammation on baseline MRI (C-score > 0.5 in at least one segment)

Exclusion Criteria:

* Prior exposure to anti-p19 biological therapy
* Exposure to more than 1 class of advanced therapies at a dose approved for the treatment of Crohn's disease (janus kinase [JAK] inhibitors, infliximab, adalimumab, certolizumab pegol, vedolizumab, ustekinumab, or approved biosimilars for these agents
* Exclude any previous use of p19 IL23s agents
* Contra-indication to mirikizumab
* Definitive ostomy
* Colectomy with IPAA
* Isolated or uncontrolled perianal lesions
* Severe obstructive symptoms
* Intra-abdominal abscess
* Contra-indication to MRI
* No health insurance
* Pregnant or lactating women
* Patients already included in biomedical research other than an observational study (e.g., registry, cohort)
* Concomitant Clostridioides difficile infection
* HIV infection
* Patient under guardianship, curatorship or safeguard of justice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Transmural response (TR25) | From week 0 to week 24
  Transmural response (TR25) define as the decrease of at least (>=) 25% of C-score in each and all active segment from baseline to week 24

SECONDARY OUTCOMES:
Clinical remission | Week 0, Week 4, Week 8, Week 12, Week 24, Week 52, Week 76
  Clinical remission will be defined according to PRO-2 (Patient Report Outcome)
Improvement or normalization of bowel urgency | Week 0, Week 4, Week 8, Week 12, Week 24, Week 52, Week 76
  Improvement or normalization of bowel urgency according to UNRS (Urgency Numerical Rating Scale)
BU clinical meaningful improvement | Week 0, Week 4, Week 8, Week 12, Week 24, Week 52, Week 76
  BU clinical meaningful improvement was defined as decrease of >=3 points; BU Remission was defined as UNRS =<2
Transmural response (TR50) | Week 0, Week 24, Week 76
  Transmural response (TR50) is defined as a decrease of at least 50% of C-score in each active segment at baseline
Transmural healing | at Week 0, Week 24, Week 76
  Transmural healing is defined as a C-score < 0.5 in each active segment at baseline
Disease activity | Week 0, Week 24, Week 76
  Disease activity is measured by the MaRIA score (Magnetic Resonance Index of activity)
IUS transmural response/healing | Week 4, Week 8, Week 12, Week 24
  IUS transmural response/healing
Bowel damage | Week 24, Week 76
  Bowel damage is measured with the Lemann Index
Transmural response (TR25) | Week 0, Week 4, Week 24, Week 76
  Transmural response will be defined as a decrease of at least 25% of C-score in each active segment at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anthony BUISSON, MD, Principal Investigator — CHU de Clermont-Ferrand; Guillaume LE COSQUER, MD, Principal Investigator — CHU de Toulouse- Hôpital Rangueil
Locations (6):
- France (6):
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest
  - CHU de Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - CHU de Nîmes Carémeau, Nîmes
  - Institut Mutualiste Monsouris, Paris
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
  - CH de Valence, Valence

IPD SHARING:
Plan to Share IPD: Undecided